CLINICAL TRIAL: NCT00473070
Title: A Clinical Study of Tobradex AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-06-37
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Drug: Tobradex AF

SUMMARY:
The purpose of this study is to determine the amount of study medication that moves from the front of the eye into the fluid at the front of the inside of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring cataract surgery

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Concentration of dexamethasone in aqueous humor following a single topical ocular administration | Periodic

SECONDARY OUTCOMES:
Changes in external and internal ocular structures, intraocular pressure, vision and other side effects | Periodic

CONTACTS AND LOCATIONS:
Overall Officials: Robert Faulkner, Study Director — Alcon Research
Locations (1):
- Pittsburgh, Pittsburgh, Pennsylvania, United States